CLINICAL TRIAL: NCT00368381
Title: A Blinded, Placebo Controlled Trial of Hydrocortisone Versus Hydrocortisone Plus Fludrocortisone for the Treatment of Adrenal Insufficiency in Severe Sepsis
Brief Title: Hydrocortisone Versus Hydrocortisone Plus Fludrocortisone for the Treatment of Adrenal Insufficiency in Severe Sepsis
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study closed for PI failure to submit renewal paperwork
Sponsor: CAMC Health System (Other)
Responsible Party: Principal Investigator, Audis Bethea, Pharm.D., Clinical Pharmacy Specialist, Trauma/Surgery, CAMC Health System
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 06-05-1813
Record Dates: First submitted 2006-08-23; First posted 2006-08-24 (Estimated); Last update posted 2012-02-13 (Estimated); Status verified 2012-02

CONDITIONS: Sepsis; Adrenal Insufficiency
Keywords: sepsis; septicemia; sepsis syndrome; adrenal insufficiency; adrenal cortex hormones; hydrocortisone; fludrocortisone
MeSH Terms: conditions — Sepsis; Adrenal Insufficiency; Systemic Inflammatory Response Syndrome | interventions — Hydrocortisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hydrocortision and fludrocortisone (Active Comparator): Study is comparing hydrocortisone alone versus the combination of hydrocortisone and fludrocortisone in the treatment of adrenal insufficiency of septic patients.
  Interventions: Drug: Hydrocortisone

INTERVENTIONS:
Drug: Hydrocortisone — Patients randomized to this arm will receive hydrocortisone for the treatment of adrenal insufficiency secondary to sepsis.

SUMMARY:
The purpose of this study is to determine if the combination of hydrocortisone plus fludrocortisone is more efficacious than hydrocortisone alone in treating adrenal insufficiency in severe sepsis.

DETAILED DESCRIPTION:
Sepsis is a significant cause of morbidity and mortality in critically ill patients in the United States. As evidenced by its increasing prevalence and high mortality rates, sepsis is a complex and difficult syndrome to treat. Current therapeutic management of sepsis includes fluid resuscitation, vasopressor and inotropic support, maintenance of oxygen delivery, drotrecogin alpha, and steroid replacement therapy in patients who are found to have adrenal insufficiency. Studies in septic patients suggest that the administration of stress doses of hydrocortisone alone, or the combination of hydrocortisone plus fludrocortisone promotes an improvement in cardiovascular performance and a quicker resolution of shock symptoms. Current therapeutic guidelines for the treatment of severe sepsis recommend either hydrocortisone alone or combination therapy with hydrocortisone and fludrocortisone as therapeutic options for the treatment of adrenal dysfunction in severe sepsis. This study will help determine which regimen is more efficacious in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Males and non-pregnant females > 18 years of age
* Patients admitted and/or pending admission to the intensive care unit
* Positive corticotropin stimulation test (Basal cortisol level of ≤ 34 μg/dL with Δ ≤ 9 μg/dL after administration of 250 mg of cosyntropin)

Patient satisfies criteria for severe sepsis Infection - one or more of the following criteria

* Documented or Suspected - positive culture results (from blood, sputum, urine, etc.)
* Anti-Infective Therapy - patient is receiving antibiotic, antifungal, or other anti-infective therapy
* Pneumonia - documentation of pneumonia (x-ray, etc.)
* WBCs - WBCs found in normally sterile .uid (urine, CSF, etc.)
* Perforated Viscus - perforation of hollow organ (bowel)

SIRS - two or more of the following

* Temperature > 38° or < 36°
* Heart rate > 90 bpm
* Respiratory rate above 20 breaths per minute
* WBC > 14,000/mm3 , < 4000/mm3, or >10% Bands

Acute organ dysfunction - one or more of the following

* Cardiovascular - SBP < 90 mmHg or MAP < 70 mmHg despite 20 mL/kg of fluid resuscitation
* Respiratory - PaO2/FiO2 ratio < 250, PEEP > 7.5, or require mechanical ventilation
* Renal - low urine output (eg, <0.5 mL/kg/hr for 1 hour despite 20mL/kg of fluid resuscitation, increased creatinine (>50% increase from baseline) or require acute dialysis
* Hematologic - low platelet count (< 100,000/mm3) or PT/PTT > upper limit of normal
* Metabolic - low pH with high lactate (eg, pH < 7.30 and plasma lactate > upper limit of normal
* Hepatic - liver enzymes > 2x upper limit of normal
* CNS - altered consciousness or reduced Glasgow Coma Score

Exclusion Criteria:

* Patients who respond to the short cosyntropin stimulation test(Δ > 9mg/dL)
* Pregnancy or breast-feeding mother
* Evidence of acute myocardial infarction, meningitis, pulmonary embolism
* AIDS (CD4 < 200 cells/mL)
* Contraindications for corticosteroids
* Formal indication for corticosteroids (specifically including patients with known adrenal insufficiency)
* Onset of shock > 24 hours
* Etomidate administration within the 6 hours preceding randomization
* Cardiac arrest prior to randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-09; Primary Completion 2009-07 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
All cause mortality | 28 days
  All cause mortality during first 28-days after study randomization.

SECONDARY OUTCOMES:
Intensive care unit survival, duration of intensive care unit stay, duration of hospitalization, survival to hospital discharge, time to vasopressor withdrawal | Unable to define
  The various secondary endpoints are patient specific serrogate markers of improvement in clinical status. Time frame for these endpoints to occur is patient specific and can not be defined for the entire study population.

CONTACTS AND LOCATIONS:
Overall Officials: John A Bethea, Pharm.D., Principal Investigator — Charleston Area Medical Center (CAMC)

REFERENCES:
- [Background] Balk RA. Severe sepsis and septic shock. Definitions, epidemiology, and clinical manifestations. Crit Care Clin. 2000 Apr;16(2):179-92. doi: 10.1016/s0749-0704(05)70106-8. PMID 10768078
- [Background] Landry DW, Oliver JA. The pathogenesis of vasodilatory shock. N Engl J Med. 2001 Aug 23;345(8):588-95. doi: 10.1056/NEJMra002709. No abstract available. PMID 11529214
- [Background] Dellinger RP. Cardiovascular management of septic shock. Crit Care Med. 2003 Mar;31(3):946-55. doi: 10.1097/01.CCM.0000057403.73299.A6. No abstract available. PMID 12627010
- [Background] Hotchkiss RS, Karl IE. The pathophysiology and treatment of sepsis. N Engl J Med. 2003 Jan 9;348(2):138-50. doi: 10.1056/NEJMra021333. No abstract available. PMID 12519925
- [Background] Vincent JL, Abraham E, Annane D, Bernard G, Rivers E, Van den Berghe G. Reducing mortality in sepsis: new directions. Crit Care. 2002 Dec;6 Suppl 3(Suppl 3):S1-18. doi: 10.1186/cc1860. Epub 2002 Dec 5. PMID 12720570
- [Background] Coursin DB, Wood KE. Corticosteroid supplementation for adrenal insufficiency. JAMA. 2002 Jan 9;287(2):236-40. doi: 10.1001/jama.287.2.236. No abstract available. PMID 11779267
- [Background] Lamberts SW, Bruining HA, de Jong FH. Corticosteroid therapy in severe illness. N Engl J Med. 1997 Oct 30;337(18):1285-92. doi: 10.1056/NEJM199710303371807. No abstract available. PMID 9345079
- [Background] Marik PE, Zaloga GP. Adrenal insufficiency in the critically ill: a new look at an old problem. Chest. 2002 Nov;122(5):1784-96. doi: 10.1378/chest.122.5.1784. PMID 12426284
- [Background] Annane D. Corticosteroids for septic shock. Crit Care Med. 2001 Jul;29(7 Suppl):S117-20. doi: 10.1097/00003246-200107001-00036. PMID 11445745
- [Background] Williamson DR, Lapointe M. The hypothalamic-pituitary-adrenal axis and low-dose glucocorticoids in the treatment of septic shock. Pharmacotherapy. 2003 Apr;23(4):514-25. doi: 10.1592/phco.23.4.514.32123. PMID 12680481
- [Background] Shenker Y, Skatrud JB. Adrenal insufficiency in critically ill patients. Am J Respir Crit Care Med. 2001 Jun;163(7):1520-3. doi: 10.1164/ajrccm.163.7.2012022. No abstract available. PMID 11401866
- [Background] Cooper MS, Stewart PM. Corticosteroid insufficiency in acutely ill patients. N Engl J Med. 2003 Feb 20;348(8):727-34. doi: 10.1056/NEJMra020529. No abstract available. PMID 12594318
- [Result] Barber AE, Coyle SM, Fischer E, Smith C, van der Poll T, Shires GT, Lowry SF. Influence of hypercortisolemia on soluble tumor necrosis factor receptor II and interleukin-1 receptor antagonist responses to endotoxin in human beings. Surgery. 1995 Aug;118(2):406-10; discussion 410-1. doi: 10.1016/s0039-6060(05)80352-6. PMID 7638758
- [Result] van der Poll T, Barber AE, Coyle SM, Lowry SF. Hypercortisolemia increases plasma interleukin-10 concentrations during human endotoxemia--a clinical research center study. J Clin Endocrinol Metab. 1996 Oct;81(10):3604-6. doi: 10.1210/jcem.81.10.8855809.
- [Result] Bone RC, Fisher CJ Jr, Clemmer TP, Slotman GJ, Metz CA, Balk RA. A controlled clinical trial of high-dose methylprednisolone in the treatment of severe sepsis and septic shock. N Engl J Med. 1987 Sep 10;317(11):653-8. doi: 10.1056/NEJM198709103171101. PMID 3306374
- [Result] Sprung CL, Caralis PV, Marcial EH, Pierce M, Gelbard MA, Long WM, Duncan RC, Tendler MD, Karpf M. The effects of high-dose corticosteroids in patients with septic shock. A prospective, controlled study. N Engl J Med. 1984 Nov 1;311(18):1137-43. doi: 10.1056/NEJM198411013111801. PMID 6384785
- [Result] Lefering R, Neugebauer EA. Steroid controversy in sepsis and septic shock: a meta-analysis. Crit Care Med. 1995 Jul;23(7):1294-303. doi: 10.1097/00003246-199507000-00021. PMID 7600840
- [Result] Cronin L, Cook DJ, Carlet J, Heyland DK, King D, Lansang MA, Fisher CJ Jr. Corticosteroid treatment for sepsis: a critical appraisal and meta-analysis of the literature. Crit Care Med. 1995 Aug;23(8):1430-9. doi: 10.1097/00003246-199508000-00019. PMID 7634816
- [Result] Thomas JP, el-Shaboury AH. Aldosterone secretion in steroid-treated patients with adrenal suppression. Lancet. 1971 Mar 27;1(7700):623-5. doi: 10.1016/s0140-6736(71)91554-6. No abstract available. PMID 4101232
- [Result] Briegel J, Forst H, Haller M, Schelling G, Kilger E, Kuprat G, Hemmer B, Hummel T, Lenhart A, Heyduck M, Stoll C, Peter K. Stress doses of hydrocortisone reverse hyperdynamic septic shock: a prospective, randomized, double-blind, single-center study. Crit Care Med. 1999 Apr;27(4):723-32. doi: 10.1097/00003246-199904000-00025. PMID 10321661
- [Result] Bollaert PE, Charpentier C, Levy B, Debouverie M, Audibert G, Larcan A. Reversal of late septic shock with supraphysiologic doses of hydrocortisone. Crit Care Med. 1998 Apr;26(4):645-50. doi: 10.1097/00003246-199804000-00010. PMID 9559600
- [Result] Annane D, Sebille V, Troche G, Raphael JC, Gajdos P, Bellissant E. A 3-level prognostic classification in septic shock based on cortisol levels and cortisol response to corticotropin. JAMA. 2000 Feb 23;283(8):1038-45. doi: 10.1001/jama.283.8.1038. PMID 10697064
- [Result] Annane D, Sebille V, Charpentier C, Bollaert PE, Francois B, Korach JM, Capellier G, Cohen Y, Azoulay E, Troche G, Chaumet-Riffaud P, Bellissant E. Effect of treatment with low doses of hydrocortisone and fludrocortisone on mortality in patients with septic shock. JAMA. 2002 Aug 21;288(7):862-71. doi: 10.1001/jama.288.7.862. PMID 12186604
- [Result] Rydvall A, Brandstrom AK, Banga R, Asplund K, Backlund U, Stegmayr BG. Plasma cortisol is often decreased in patients treated in an intensive care unit. Intensive Care Med. 2000 May;26(5):545-51. doi: 10.1007/s001340051202. PMID 10923728
- [Result] Oelkers W. Adrenal insufficiency. N Engl J Med. 1996 Oct 17;335(16):1206-12. doi: 10.1056/NEJM199610173351607. No abstract available. PMID 8815944
- [Result] Zipser RD, Davenport MW, Martin KL, Tuck ML, Warner NE, Swinney RR, Davis CL, Horton R. Hyperreninemic hypoaldosteronism in the critically ill: a new entity. J Clin Endocrinol Metab. 1981 Oct;53(4):867-73. doi: 10.1210/jcem-53-4-867. PMID 6270176
- [Result] Findling JW, Waters VO, Raff H. The dissociation of renin and aldosterone during critical illness. J Clin Endocrinol Metab. 1987 Mar;64(3):592-5. doi: 10.1210/jcem-64-3-592. PMID 3029157